CLINICAL TRIAL: NCT00619606
Title: A Randomised, Parallel, Open Label Study to Determine the Efficacy of a New Oral-Nasal Oxygenating Device (TwinGuard) Compared to Standard Bite Block Plus Nasal Cannulae
Brief Title: To Determine the Efficacy of the TwinGuard in Oxygen Delivery During and Post Endoscopic Procedure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trawax Pty Limited (Other)
Responsible Party: Julie Nunn, Trawax Pty Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDD05/C05; TGA CTN 089/2006
Record Dates: First submitted 2008-01-31; First posted 2008-02-21 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Hypoxia; Hypercapnia
Keywords: prevention of hypoxia; prevention of hypercapnia
MeSH Terms: conditions — Hypoxia; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: TwinGuard — A system consisting of an endoscopic bite block that fits together with a nasal cannula. After gastroscopy, the bite block is discarded leaving the patient receiving oxygen in recovery.An optional carbon dioxide sampling device fits with the TwinGuard in endoscopy to monitor expired air.
Device: Standard endoscopic bite block — Placed in the mouth during gastroscopy to protect the endoscope and the patient's teeth
Device: Standard nasal cannula — Delivers oxygen to the nose. Tubing runs from the nose around the back of the ears and under the chin which then runs to an oxygen source.
Device: CO2 sample line — Samples expired air from a patients nose. Tubing is connected to a capnograph.

SUMMARY:
A comparative study which compares the end-tidal carbon dioxide and oxygen saturation levels of patients during endoscopy which have used either the new oral-nasal oxygenating device (TwinGuard), or a standard bite block plus nasal cannulae using an equivalent flow rate of oxygen.

DETAILED DESCRIPTION:
Hypoxia is common during endoscopy. Following sedation induction, oxygen saturation falls moderately in most patients, whilst some drop to unacceptable levels. To monitor such changes endoscopic practices routinely use oximeters and capnography.

TwinGuard is an all-in-one device which incorporates a bite block with the functionality of nasal cannula as well as monitoring expired air (carbon dioxide)

ELIGIBILITY:
Inclusion Criteria:

* Provided written fully informed consent as per protocol
* No clinical evidence of significant respiratory conditions
* Fasted for 6 hours prior to enrolment as per standard clinical practice for panendoscopy

Exclusion Criteria:

* Patients suffering from cardio respiratory disease, moderate to severe asthma, lung and heart disease
* Patients who have a history of drug or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Borody, Principal Investigator — Centre for Digestive Diseases, Sydney